CLINICAL TRIAL: NCT05183308
Title: The Effect of Combined Drug Therapy in Lateral Fragility Fractures of the Femur:a Clinical Study
Brief Title: Combined Drug Therapy in Lateral Fragility Fractures of the Femur
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari (Other)
Responsible Party: Sponsor
Other Study IDs: Femur-Clodronic Acid
Record Dates: First submitted 2021-12-21; First posted 2022-01-10 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2020-12

CONDITIONS: Femur Fracture
Keywords: fragility lateral femoral fractures; bisphosphonates; clodronic acid; bone density
MeSH Terms: conditions — Femoral Fractures | interventions — Clodronic Acid

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients treated with Vitamin D
- patients treated with Vitamin D and Clodronic Acid
  Interventions: Drug: Clodronic Acid

INTERVENTIONS:
Drug: Clodronic Acid — Osteoporotic fracture treated with surgical and medical therapy
  Groups: patients treated with Vitamin D and Clodronic Acid

SUMMARY:
It was conducted a prospective study with a series of 50 patients treated by intramedullary nail using Clodronic acid and Vitamin D (study group including 25 patients) and patients with the same fractures treated with Vitamin D alone (control group including 25 patients).

One independent observer performed clinical, biochemical and functional evaluations at T0 (1st day post-surgery) and at T1 (12 months later) Biochemical markers (serum calcium level, serum phosphate level, PTH (parathormone), Vitamin D, serum C-terminal telopeptide), VAS (Visual Analogic Scale) and HHS (Harris Hip Score) score, and femur densitometric views were administered at each evaluation.

ELIGIBILITY:
Inclusion Criteria:

* femur fractures type 31-A1, A2, (Muller ME, Nazarian S, Kock P et al.);
* age 60 - 85 years;
* co-operative patients;
* Body Mass Index (BMI) < 30 Kg/m²;
* patients treated by intramedullary nailing surgery (PFNA Synthes®);
* patients with osteoporosis disease if T-Score< -2,5;

Exclusion Criteria:

* patients with heart, kidney, neurological diseases;
* patients with metabolic and systemic disease (rheumatoid arthritis, diabetes mellitus);
* previous surgery or severe osteoarthritis of lower limbs;
* specific drugs treatments such as anticoagulants or psychiatric drugs.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Fifty (50) patients referring to the Orthopaedic and Trauma Unit of the local University Hospital between May 2019 and March 2020 with lateral fragility fracture were prospectively recruited.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Change in Visual Analogic Scale | Day 1; Month 12 (after surgey)
  The Hip Pain was quantified using the Visual Analogic Scale ranging between 0 (no pain) and 10 points (worst imaginable pain).

CONTACTS AND LOCATIONS:
Locations (1):
- AOUC Policlinico di Bari - UOC Ortopedia e Traumatologia, Bari, Italy

IPD SHARING:
Plan to Share IPD: No